CLINICAL TRIAL: NCT07136298
Title: Seizure Semiology Identification and Agreement in the Intensive Care Setting: How do Clinical Scientists Compare to Other Healthcare Professionals (Intensivists, Neurologists, ITU Nurses and Neurophysiologists) in Identifying and Interpreting Clinical Signs in Patients on the Adult Intensive Care Unit
Brief Title: Seizure Identification on the Intensive Care Unit (ICU)
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24CN001
Record Dates: First submitted 2025-07-18; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Seizures
Keywords: Intensive Care; Clinical Scientist; Neurologists; Intensivists; ITU Nurses
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Clinical Scientists
  Interventions: Other: Clinical Opinion
- Advanced Clinical Practitioners
  Interventions: Other: Clinical Opinion
- Intensivists
  Interventions: Other: Clinical Opinion
- Clinical Neurophysiologists
  Interventions: Other: Clinical Opinion
- Neurologists
  Interventions: Other: Clinical Opinion
- ICU Nurses
  Interventions: Other: Clinical Opinion

INTERVENTIONS:
Other: Clinical Opinion — Staff participants will be asked to review video clips of events captured during EEGs performed on the ICU and asked to state whether they think the event was an epileptic seizure or not, and what aspects of each event led them to that decision

SUMMARY:
The aim of this project is to assess the ability of different groups of National Heath Service (NHS) professionals to correctly identify clinical seizures, and distinguish them from other movements commonly seen in the ICU environment, when shown digital video recordings only.

Patients on the ICU are at risk of having seizures, however also commonly make other movements, including shivering, jerking, tics and tremors. An Electroencephalogram (EEG) records the brain wave activity and can help distinguish epileptic seizures from other movements. In a study by Bendadis et al (2010), 52 video-EEGs were reviewed containing "possible seizures" on the ICU. They found only 27% recorded actual epileptic events, with the other 73% having a range of other movements. Malone et al (2009) studied accuracy of diagnosis of 20 video recordings of clinical episodes on the neonatal unit, comparing different staff groups. They found no significant difference between Doctors and Nurses in correctly identifying seizures, however found that accuracy of diagnosis was generally poor.

Clinical scientists are currently expanding their roles and responsibilities across Neurophysiology, including giving consultant-level advice on EEG investigations. EEG recordings on the ICU are often obscured by excessive, unavoidable electrical/movement artefacts caused by equipment such ventilators and pumps, and patient factors such as position, breathing artefact and suctioning. These make the EEG difficult to interpret (Boggs 2021). Assessing the clinical signs and symptoms which we may see in ICU patients, in the absence of interpretable EEG, is an essential skill.

This study aims to assess Clinical Scientists skills at clinical interpretation, in comparison with other staff groups in the ICU setting. Staff will be asked to watch video clips of events captured in the ICU, and tell us whether they think they are seizures or not, and explain their thought process behind the decision.

ELIGIBILITY:
Inclusion Criteria:

Staff working at Nottingham University Hospitals (NUH) in one of the following staff groups;

* Neurophysiology Scientists/Clinical Physiologists at Band 7 level and above,
* Neurophysiologists who have completed the CCT in Neurophysiology with at least 1 year of Adult ICU experience.
* members of the Neurology medical team with at least 1 years' experience of covering ITU
* Intensivists with at least 1 year's experience working on the Adult intensive care unit
* Nursing staff working on the Intensive care unit with at least 1 year's experience

Exclusion Criteria:

* Staff not employed by NUH i.e. agency staff
* Staff in other groups not mentioned above

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population are staff working in the Adult ICU at Nottingham University Hospitals, in one of the following groups; Neurophysiology Scientists/Clinical Physiologists, Neurophysiologists, Neurologists, Intensivists, Advanced Clinical Practitioners and Nursing Staff
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Level of Agreement | through study completion, an average of 1 year
  The primary outcome measure is the level of agreement between the clinical opinion of the different staff groups and the EEG result

SECONDARY OUTCOMES:
Interrater Reliability | through study completion, an average of 1 year
  The level of agreement between the different individuals in each staff group.
Thematic Analysis | through study completion, an average of 1 year
  thematic analysis of the decision making process (based on the free text justifications for why individuals made the choice they did)

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals, Nottingham, Nottinghamshire, United Kingdom